CLINICAL TRIAL: NCT06738654
Title: Application of Single-Port Robot-Assisted Breast-Conserving Surgery Via Axillary Approach for Breast Cancer.
Acronym: 单孔机器人-SPR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Yan (Other)
Responsible Party: Sponsor-Investigator, Xu Yan, Yan Xu,MD., PhD. Department of Breast and Thyroid Surgery Daping Hospital, Army Medical University, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCIIT241104
Record Dates: First submitted 2024-11-29; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Invasive Breast Carcinoma
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Experimental Group: Breast-conserving surgery for breast cancer using single-port robotic surgery.
  Control Group: Breast-conserving surgery for breast cancer using traditional open surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Breast-conserving surgery for breast cancer using traditional open surgery.
  Interventions: Procedure: traditional open surgry
- Experimental Group (Experimental): Breast-conserving surgery for breast cancer using single-port robotic surgery.
  Interventions: Procedure: robot-surgery

INTERVENTIONS:
Procedure: robot-surgery — Breast-conserving surgery for breast cancer using single-port robotic surgery.
  Arms: Experimental Group
Procedure: traditional open surgry — Breast-conserving surgery for breast cancer using traditional open surgery.
  Arms: Control Group

SUMMARY:
Evaluate the safety and feasibility of single-port robotic surgery in breast-conserving surgery, compare and analyze the advantages and disadvantages of single-port robotic surgery and open surgery in terms of complications, postoperative complications, perioperative recovery effects, and safety in breast cancer breast-conserving surgery, in order to select a more effective and safe surgical method. Subjects who meet the inclusion criteria will enter the research process, with surgery including SPr-breast-conserving surgery or open-breast-conserving surgery, and the choice of the two surgical methods is based on the patient's financial situation and the availability of equipment;

DETAILED DESCRIPTION:
Evaluate the safety and feasibility of single-port robotic surgery in breast-conserving surgery, compare and analyze the advantages and disadvantages of single-port robotic surgery and open surgery in terms of complications, postoperative complications, perioperative recovery effects, and safety in breast cancer breast-conserving surgery, in order to select a more effective and safe surgical method. Subjects who meet the inclusion criteria will enter the research process, with surgery including SPr-breast-conserving surgery or open-breast-conserving surgery, and the choice of the two surgical methods is based on the patient's financial situation and the availability of equipment; - Preoperative hospitalization period: Collect patient disease information (including mammography, breast ultrasound, breast enhanced MRI, etc.) - On the day of surgery: Record operating time, intraoperative blood loss, intraoperative complications, intraoperative adverse events, etc.; - Postoperative hospitalization period: Record postoperative complications (postoperative bleeding, necrosis of the flap or nipple-areola complex, subcutaneous emphysema, infection, capsule spasm, postoperative shoulder pain and discomfort, etc.), postoperative pain scores, postoperative pathological biopsy; - Postoperative hospital stay: Calculated from the day of surgery to the day of discharge; - 28 days postoperatively: Understand the complication rate and mortality rate within 28 days postoperatively; - 90 days postoperatively: Understand the complication rate and mortality rate within 90 days postoperatively; - 3-year disease-free survival period (calculated from the time of surgery to the last follow-up or recurrence and metastasis date, recurrence is defined as recurrence in the surgical area and distant metastasis); - 3-year overall survival rate (calculated from the time of surgery to the last follow-up or death).

ELIGIBILITY:
Inclusion Criteria:

1. The patient himself has very high requirements for beauty, and requires no scar on the chest;
2. No chest surgery and radiotherapy.
3. No contraindications to surgery and anesthesia.
4. Clinical I, stage of early breast cancer and the breast has an appropriate volume, can maintain a good breast shape after surgery.
5. Patients in the clinical period who meet the standard of breast conservation surgery after preoperative treatment.
6. Age: 18 and 65 years old.

Exclusion Criteria:

1. Inflammatory breast cancer.
2. The tumor is extensive and it's difficult to achieve negative margins or an ideal breast - conserving appearance.
3. Diffusely distributed malignant - characteristic calcifications.
4. The margin is positive after local extensive tumor resection, and a negative margin in pathological examination still can't be ensured after re - resection.
5. The patient refuses.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The successful rate of breast-conserving surgery | From enrollment to the end of treatment at 2 weeks
  Whether intraoperative frozen section biopsy of the surgical margins detects cancer cells; if it is negative after two or fewer attempts, then the breast-conserving surgery is considered successful.

CONTACTS AND LOCATIONS:
Locations (1):
- Aramy medical center., Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
it contains privacy about patients

REFERENCES:
- [Derived] Yu F, Zhang G, Guo L, Luo F, Chen Y, Xu Y. Single-Port Robotic-assisted Transaxillary Breast-conserving Surgery: A Prospective, Single-arm, Non-randomized Phase IIa Clinical Trial. J Vis Exp. 2025 Aug 19;(222). doi: 10.3791/68459. PMID 40920680

DOCUMENTS (2):
  • Statistical Analysis Plan (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT06738654/SAP_000.pdf
  • Informed Consent Form (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT06738654/ICF_001.pdf